CLINICAL TRIAL: NCT00361153
Title: Effects on Colesevelam HC1 (WelChol®) on Insulin Sensitivity in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Vice President Clinical Development, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WEL-202
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Colesevelam hydrochloride
  Interventions: Drug: Colesevelam hydrochloride
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Colesevelam hydrochloride — Welchol tablet 625mg
  Other Names: Welchol
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This study is designed to test whether WelChol (colesevelam HC1) improves blood sugar control in patients with type 2 diabetes by making their own insulin work more efficiently.

DETAILED DESCRIPTION:
Single-center, randomized, parallel, double-blind, placebo controlled, 8-week trial in subjects with type 2 diabetes mellitus. Two parallel treatment groups include double-blind colesevelam or placebo. A screening period may be up to 18 weeks to withdraw non sulfonylurea antidiabetic treatment or withdraw or adjust sulfonylurea antidiabetic treatment. To evaluate hepatic and peripheral insulin sensitivity, subjects will undergo a two-step hyperinsulinemic-euglycemic clamp with a tritiated glucose infusion at pre randomization and after 8 weeks of treatment. To evaluate oral glucose absorption, subjects will undergo two oral glucose tolerance tests (OGTT) at pre randomization, one without colesevelam and one with colesevelam, and one OGTT at the end of the treatment period..

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria at the Screening Visit will be eligible to participate in the trial:

* Have given written informed consent
* Ages 18 to 75 years, inclusive
* Diagnosis of type 2 diabetes mellitus of at least 3 months duration
* HbA1C 7.0- 10.0%, inclusive
* Antidiabetic treatment may include oral agents; all antidiabetic agents must be withdrawn before randomization
* Women may be enrolled if they are not pregnant (negative serum βHCG at the Screening Visit), are not breast-feeding, and do not plan to become pregnant during the trial. In addition, they must either have had a hysterectomy or tubal ligation at least 6 months before signing informed consent, be post-menopausal for 1 year, or practicing an acceptable method of birth control. An acceptable method of birth control may be oral, injectable or implantable hormonal contraceptives, intrauterine device, diaphragm plus spermicide, or female condom plus spermicide. Abstinence, partner's use of condoms, and partner's vasectomy are NOT acceptable methods of contraception
* BMI 25 - 45 kg/M sq, inclusive

Exclusion Criteria:

Subjects are excluded from participation in the study if any of the following criteria apply:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Treatment with lipid or blood pressure lowering therapy that has not been stable for three months before randomization
* Treatment with WelChol, cholestyramine or colestipol for hyperlipidemia within the last 3 months
* Treatment with thiazolidinediones
* History of dysphagia, swallowing disorders, or intestinal motility disorder
* Serum triglyceride >500 mg/dL at Visit 1
* Serum LDL-C <60 mg/dL at Visit 1
* Any condition or therapy which, in the opinion of the investigator, poses a risk to the subject or makes participation not in the subject's best interest
* Use of any investigational drug within 30 days before randomization
* Chronic treatment with oral corticosteroids
* History of hyperthyroidism and/or treatment with thyroid hormone/ levothyroxine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of 8 weeks treatment with WelChol on insulin sensitivity,as measured by the hyperinsulinemic-euglycemic clamp method, i.e., placebo-corrected change from baseline in M-value. | 8 weeks

SECONDARY OUTCOMES:
To evaluate the effect of 2 weeks treatment with WelChol on insulin sensitivity,as measured by the hyperinsulinemic-euglycemic clamp method. | 2 weeks
To evaluate acute and chronic effects of treatment with WelChol on plasma glucose after ingestion of a standard meal replacement. | 8 weeks
To evaluate the effect of treatment with WelChol on HbA1C, insulin, fasting plasma glucose, and fructosamine. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Development, Study Director — Daiichi Sankyo
Locations (1):
- Diabetes and Glandular Research Associates, San Antonio, Texas, United States

REFERENCES:
- [Derived] Schwartz SL, Lai YL, Xu J, Abby SL, Misir S, Jones MR, Nagendran S. The effect of colesevelam hydrochloride on insulin sensitivity and secretion in patients with type 2 diabetes: a pilot study. Metab Syndr Relat Disord. 2010 Apr;8(2):179-88. doi: 10.1089/met.2009.0049. PMID 20059361